CLINICAL TRIAL: NCT00452205
Title: Bone Marrow-derived Cells' Contribution to Tumor Formation and Epithelial Cells Regeneration in the Gastrointestinal Tract
Brief Title: Bone Marrow-derived Cells' Contribution to Tumor Formation and Inflammation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Komagome Hospital (Other)
Responsible Party: Naoto Egawa, Tokyo Metropolitan Komagome Hospital
Other Study IDs: CICK-07521
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Gastrointestinal Neoplasms
Keywords: bone marrow-derived stem cell; bone marrow transplantation; graft versus host disease; gastrointestinal cancer; after receiving bone marrow transplantation
MeSH Terms: conditions — Gastrointestinal Neoplasms; Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to clarify the relationship bone marrow-derived cells and the formation of the tumors, and the role of these cells in regeneration of epithelial cells in the gastrointestinal tract.

DETAILED DESCRIPTION:
Recent experimental studies showed that circulating bone marrow-derived stem cells contribute to the formation of cancers cells. However, it is not clear whether this is applicable to human beings or not. In addition, bone marrow-derived cells are considered to play a significant role in regeneration of inflamed epithelial cells of the gastrointestinal tract during graft versus host disease (GVHD), which sometimes occurs after bone marrow transplantation (BMT). On the other hand, it is well known that the incidence of solid tumors is significantly increased following bone marrow transplantation.

One purpose of this study is to determine the role of bone marrow-derived cells in the tumor formation and acute or chronic inflammation of the gastrointestinal tract in human beings, and the other is to discover early cancers of the gastrointestinal tract in the subjects received BMT by conducting surveillance for detecting second tumor, periodically.

All subjects are the patients received allogeneic BMT in Tokyo Metropolitan Komagome Hospital for hematopoietic disorders.

For determining the role of bone marrow-derived cells in the solid tumors and inflammation like GVHD, suitable candidates are females who received allogeneic BMT from male donors, because the most reliable marker of bone marrow-derived cells is identification of the Y chromosomes from the male donor in the tissue of female.

For the early detection of gastrointestinal cancers, the subjects are confined to patients without recurrence of original disorder at least 1 year after BMT. They are scheduled to undergo a medical inspection using gastrointestinal endoscopy, periodically.

When tumor or any other lesions are discovered, biopsy specimens are taken and proceed to pathological examination. According to the results, the patients will have proper treatments.

The tissue specimens from the tumors or inflammation in female recipients from male donors are processed for Y fluorescent in situ hybridization (FISH) analysis and immunocytochemistry using monoclonal antibodies such as cytokeratin, CD45 and so on.

Procedure

First of all, informed consent to this study should be gained from the subjects.

Study 1: to determine the role of bone marrow-derived cells on inflammation such as GVHD

1. Subjects are female recipients from male donors.
2. When they have some symptoms suggesting acute or chronic GVHD, gastrointestinal endoscopy is conducted and biopsy specimens are taken from the lesions for the definite diagnosis and identification of bone marrow-derived cells.
3. Pathological investigation(Y-FISH etc.) is conducted using the tissue specimens.

Study 2: to conduct surveillance for second malignancy and to determine the role of bone marrow-derived cells on the formation of the tumor

1. Subjects are confined to bone marrow recipients without the recurrence of the original disorder at least 1 year after BMT.
2. A medical inspection for gastrointestinal tract is performed using periodical endoscopy.
3. The tissue from tumors or any other lesions discovered are taken as biopsy specimen and processed for pathological examination. Regarding the female recipients from male donors, the same procedure as in the study 1 is taken for pathological study.

ELIGIBILITY:
Inclusion Criteria:

* After allogeneic bone marrow transplantation

Exclusion Criteria:

* Contraindication for gastrointestinal endoscopy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients received bone marrow transplantation in Tokyo Metropolitan Komagome Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-04; Study Completion 2017-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Egawa, MD, Study Director
Locations (1):
- Cancer and Infection Disease Center, Komagome, Tokyo, Bunkyo-ku, Japan

REFERENCES:
- [Background] Houghton J, Stoicov C, Nomura S, Rogers AB, Carlson J, Li H, Cai X, Fox JG, Goldenring JR, Wang TC. Gastric cancer originating from bone marrow-derived cells. Science. 2004 Nov 26;306(5701):1568-71. doi: 10.1126/science.1099513. PMID 15567866